CLINICAL TRIAL: NCT01891422
Title: Longitudinal Studies of the Glycoproteinoses
Status: Completed | Type: Observational
Sponsor: Greenwood Genetic Center (Other)
Responsible Party: Sponsor
Other Study IDs: GGC75
Record Dates: First submitted 2013-05-22; First posted 2013-07-03 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Aspartylglucosaminuria; Fucosidosis; Galactosialidosis; Alpha Mannosidosis; Beta Mannosidosis; Mucolipidosis II; Mucolipidosis III; Schindler Disease; Sialidosis
Keywords: Glycoprotein Storage Disease; Lysosomal Storage Disease; mannosidase deficiency disorders; Neuraminidase deficiency with beta-galactosidase deficiency; mucolipidoses; Oligosaccharidoses; Lysosomal Disease; Metabolic Disease, Inborn; aspartylglucosaminuria; fucosidosis; galactosialidosis; alpha mannosidosis; beta mannosidosis; mucolipidosis II; mucolipidosis III; Schindler disease; sialidosis
MeSH Terms: conditions — Aspartylglucosaminuria; Fucosidosis; Neuraminidase deficiency with beta-galactosidase deficiency; alpha-Mannosidosis; beta-Mannosidosis; Mucolipidoses; Schindler Disease, Type I; Glycoprotein Storage Disease; Lysosomal Storage Diseases; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — When applicable, plasma, white cells, fibroblasts, urine.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Non-interventional.

SUMMARY:
The glycoproteinoses are among the most rare and least researched of the lysosomal diseases. The diseases include aspartylglucosaminuria, fucosidosis, galactosialidosis, alpha-mannosidosis, beta-mannosidosis, mucolipidosis II, mucolipidosis III, Schindler disease, and sialidosis. Longitudinal studies of these conditions are needed in order to better define how common the diseases are, identify clinical features which could contribute to early diagnoses, detail progression of the diseases, assess the supportive therapies currently used, and identify potential treatments. Laboratory tests will evaluate metabolic and genetic defects found in participants' blood and urine samples.

DETAILED DESCRIPTION:
This is a longitudinal study of 100 individuals diagnosed with any one of the nine glycoproteinoses. Because of the small number of individuals diagnosed with these diseases, participants will be strongly encouraged to be evaluated in person at a study site, but inability to travel to a study site will not exclude a person from participating. This non-interventional study will also collect medical information about participants through questionnaire, phone interviews, and review of medical records regarding the person's usual medical care, including lab testing and x-rays or other imaging studies.

Participants who are evaluated at the study center will have a physical examination performed by a clinical geneticist and neuropsychological studies administered by the study psychologist. Neuropsychological studies assess intelligence, learning abilities, language skills, and ability to participate in day to day activities of life. Participants seen at the study center will have skeletal x-rays performed to evaluate the impact of the disease on the participant's bones.

Every participant will complete (or have a care provider complete for them)

* A questionnaire about their birth, development, and medical history
* An interview with study personnel (in person or via telephone)
* Follow up interviews on at least an annual basis to update the medical history

Each participant will be asked to

* Give a blood sample
* Give a urine sample
* Some participants may be asked to give a skin biopsy.

ELIGIBILITY:
Inclusion Criteria:

Be an individual of any age diagnosed with one of the following conditions

* Aspartylglucosaminuria
* Fucosidosis
* Galactosialidosis
* alpha mannosidosis
* beta mannosidosis
* Mucolipidosis II
* Mucolipidosis III
* Schindler disease
* Sialidosis

Exclusion Criteria:

* not diagnosed with one of the nine glycoproteinoses listed above.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals of any age diagnosed with any of the nine glycoproteinoses will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-08; Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Change in Disease Characteristics Over Time | Baseline, Year 1, Year 2, Year 3, Year 4
  Specific characteristics will be assessed by history and medical record review, to include: onset of disease presentation (signs and symptoms); age at presentation; timeframe of developmental milestones; milestones for educational achievement and cognitive measures; surgical procedures- when performed and outcomes; growth data over time; and indications for subspecialist care (for example cardiology, orthopedics, neurology).

SECONDARY OUTCOMES:
Identification of Genotype-Phenotype Correlation | Baseline
  Molecular and biochemical tests will be performed at subjects' baseline visits to confirm disease identity, and to identify genotype-phenotype correlations.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Cathey, MD, Principal Investigator — Greenwood Genetic Center
Locations (1):
- Greenwood Genetic Center, North Charleston, South Carolina, United States

REFERENCES:
- [Background] Kerr DA, Memoli VA, Cathey SS, Harris BT. Mucolipidosis type III alpha/beta: the first characterization of this rare disease by autopsy. Arch Pathol Lab Med. 2011 Apr;135(4):503-10. doi: 10.5858/2010-0236-CR.1. PMID 21466370
- [Background] David-Vizcarra G, Briody J, Ault J, Fietz M, Fletcher J, Savarirayan R, Wilson M, McGill J, Edwards M, Munns C, Alcausin M, Cathey S, Sillence D. The natural history and osteodystrophy of mucolipidosis types II and III. J Paediatr Child Health. 2010 Jun;46(6):316-22. doi: 10.1111/j.1440-1754.2010.01715.x. Epub 2010 Mar 29. PMID 20367762
- [Result] Cathey SS, Leroy JG, Wood T, Eaves K, Simensen RJ, Kudo M, Stevenson RE, Friez MJ. Phenotype and genotype in mucolipidoses II and III alpha/beta: a study of 61 probands. J Med Genet. 2010 Jan;47(1):38-48. doi: 10.1136/jmg.2009.067736. Epub 2009 Jul 16. PMID 19617216
- See also: Greenwood Genetic Center — http://www.ggc.org